CLINICAL TRIAL: NCT02783170
Title: A Prospective, Randomized, Open-label Clinical Trial to Assess the Safety and Immunogenicity of Simultaneous vs Sequential Administration of Tetanus Toxoid, Reduced Diphtheria Toxoid, and Acellular Pertussis Vaccine and Inactivated Influenza Vaccine in Pregnant Women - Pilot
Brief Title: Safety and Immunogenicity of Simultaneous Tdap and IIV in Pregnant Women
Acronym: Tdap/IIV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00071192
Record Dates: First submitted 2016-05-11; First posted 2016-05-26 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2019-05

CONDITIONS: Pregnancy
Keywords: Tdap vaccine; Flu vaccine; vaccines in pregnancy; immunizations in pregnancy; Whooping Cough; Pertussis; Influenza
MeSH Terms: conditions — Influenza, Human; Whooping Cough | interventions — Diphtheria-Tetanus-Pertussis Vaccine; Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simultaneous vaccination arm (Other): In the study arm,subjects will receive both Tdap and IIV vaccines during study visit 1.
  Interventions: Biological: Tetanus, Diphtheria, and Pertussis Vaccine; Biological: 2016-2017 Quadrivalent Inactivated Influenza Vaccine; Biological: 2017-2018 Quadrivalent Inactivated Influenza Vaccine
- Sequential vaccination arm (Other): In this study arm, subjects will receive the IIV vaccine during study visit 1. Approximately 3 weeks later, they will receive the Tdap vaccine during study visit 4.
  Interventions: Biological: Tetanus, Diphtheria, and Pertussis Vaccine; Biological: 2016-2017 Quadrivalent Inactivated Influenza Vaccine; Biological: 2017-2018 Quadrivalent Inactivated Influenza Vaccine

INTERVENTIONS:
Biological: Tetanus, Diphtheria, and Pertussis Vaccine
  Other Names: Tdap
Biological: 2016-2017 Quadrivalent Inactivated Influenza Vaccine
  Other Names: Flu vaccine; 2016-2017 Flu vaccine
Biological: 2017-2018 Quadrivalent Inactivated Influenza Vaccine
  Other Names: Flu vaccine; 2017-2018 Flu vaccine

SUMMARY:
This is a pilot, prospective, randomized, open-label clinical trial. During the study, pregnant women will be randomized (1:1) to receive co-administration of a single intramuscular (IM) 0.5 mL dose of US-licensed inactivated influenza vaccine (IIV) and a single intramuscular (IM) 0.5 mL dose of US-licensed Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine adsorbed (Tdap) or sequential administration of the vaccines (IIV followed by Tdap ~ 21 days later). Vaccines will be administered by licensed study personnel.

Prior Tdap/Td/TT and influenza vaccine history will be verified by medical record review when possible.

Injection-site (local) and systemic reaction data will be assessed on vaccination day and during the 7 days following vaccination using either identical web-based or paper diaries, depending on study participant preference.

Maternal serum samples will be collected for antibody titers relevant to the Tdap and Influenza at time points that include: prior to vaccination(s), ~21 days post vaccination(s), and at delivery. Additionally, cord blood serum will be analyzed for the same antibody titers.

Pregnant women will be followed with comprehensive obstetric and neonatal outcomes obtained from medical record review.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant, as determined by medical history; 18 - 45 years of age inclusive
2. Intention of receiving Tdap and IIV vaccines based on Advisory Committee on Immunization Practices (ACIP) recommendations
3. Willing to provide written informed consent prior to initiation of any study procedures
4. Singleton gestation ≥ 26 weeks 0 days gestation - ≤32 weeks 0 days gestation at the time of Visit 1 vaccination based on reconciliation of last menstrual period and ultrasound dating. Estimated due date (EDD) and Gestational Age (GA) - EDD will be based on reconciliation of a "sure" first day of the last menstrual period (LMP) and earliest dating ultrasound. If the LMP is uncertain, then the earliest dating ultrasound will be used to determine EDD and GA. If the ultrasound derived-EDD is in agreement with sure-LMP derived EDD, then the LMP-derived EDD is used to determine GA. If the ultrasound derived EDD is not in agreement with the LMP-derived EDD, the ultrasound-derived EDD is used to determine GA.
5. English or Spanish literate
6. Intention of being available for entire study period and complete all relevant study procedures, including follow-up phone calls and collection of delivery information.

Exclusion Criteria:

1. For subjects enrolling during the 2016-2017 influenza season: IIV/LAIV receipt during 2016-2017 influenza season prior to study enrollment
2. For subjects enrolling during the 2017-2018 influenza season: IIV/LAIV receipt during 2017-2018 influenza season prior to study enrollment

   2. Tdap/Td/TT receipt during current pregnancy prior to study enrollment 3. Has immunosuppression as a result of an underlying illness or treatment, or use of anti-cancer chemotherapy or radiation therapy within the preceding 36 months.

   4. Has an active neoplastic disease (excluding non-melanoma skin cancer), a history of any hematologic malignancy, current bleeding disorder, or taking anticoagulants (daily low dose aspirin may be acceptable).

   5. Has a history of receiving immunoglobulin or other blood product (with exception of Rhogam) within the 3 months prior to enrollment in this study.

   6. Known to have pre-existing diabetes mellitus or an autoimmune disorder. 7. Febrile illness within the last 24 hours or an oral temperature >/= 100.4°F (>/= 38.0°C) prior to IIV or Tdap administration 8. Contraindication to IIV receipt including history of severe allergic reaction after a previous dose of any influenza vaccine; or to a vaccine component, including egg protein 9. Contraindication to Tdap receipt including history of severe allergic reaction after a previous dose of any tetanus toxoid-, diphtheria toxoid-, or pertussis antigen-containing vaccine or encephalopathy within 7 days of administration of a previous dose of a pertussis antigen-containing vaccine that is not attributable to another identifiable cause 10. Arthus-type hypersensitivity reaction following a prior dose of a tetanus toxoid-containing vaccine within the last 10 years 11. Any condition that may interfere with assessment of local injection site reactions, e.g. lymphadenectomy or obscuring tattoos 12. History of Guillain-Barré syndrome within 6 weeks of a prior dose of any tetanus toxoid-, diphtheria toxoid- or pertussis antigen-containing vaccine or influenza vaccine 13. Known or suspected impairment of immunologic function including infection with HIV, hepatitis B or C 14. Use of immunosuppressive or cytotoxic drugs except receipt of oral or parenteral (intravenous, subcutaneous or intramuscular) corticosteroids 30 or more days prior to enrollment. Persons who have used oral or parenteral corticosteroids within 12 months prior to enrollment may be enrolled if the longest course of therapy was less than 14 consecutive days and no dose was given within 30 days of enrollment. Intraarticular, bursal, tendon, or epidural injections of corticosteroids are permissible if the most recent injection was 30 or more days prior to enrolment. Persons applying topically corticosteroid in either upper arm (i.e. injection site) may be enrolled 1 or more days after their therapy is completed. Corticosteroids administered topically at non-injection sites, by inhalation or intranasally are permissible 15. Receipt of any licensed vaccine within 14 days prior to study vaccination or planning receipt of any vaccines (except study vaccines) prior to Visit 7 follow up.

   16. Receipt of live vaccine during current pregnancy. 17. High risk for preterm birth (active preterm labor, short cervix, cervical cerclage, receipt of antenatal corticosteroids for fetal lung maturity prior to Visit 1) 18. Antenatal ultrasound diagnosis of fetal growth restriction, defined as < 10th percentile estimated fetal weight for gestational age 19. Known fetal congenital anomaly, e.g. genetic abnormality or malformation based on antenatal ultrasound 20. Any condition which, in the opinion of the investigators, may pose a health risk to the subject or interfere with the evaluation of the study objectives.

   21. Anyone who is a relative of any research study personnel 22. Anyone who is an employee of any research study personnel 23. Anyone who is already enrolled or plans to enroll in another clinical trial with an investigational product. Co-enrollment in observational or behavioral intervention studies are allowed at any time.

   24. Previous participation in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2016-09; Primary Completion 2018-04-03 (Actual); Study Completion 2018-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geeta Swamy, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Centers for Disease Control and Prevention, Atlanta, Georgia
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Simultaneous Vaccination Arm: In the study arm,subjects will receive both Tdap and IIV vaccines during study visit 1.
  Tetanus, Diphtheria, and Pertussis Vaccine
  2016-2017 Quadrivalent Inactivated Influenza Vaccine
  2017-2018 Quadrivalent Inactivated Influenza Vaccine
- Sequential Vaccination Arm: In this study arm, subjects will receive the IIV vaccine during study visit 1. Approximately 3 weeks later, they will receive the Tdap vaccine during study visit 4.
  Tetanus, Diphtheria, and Pertussis Vaccine
  2016-2017 Quadrivalent Inactivated Influenza Vaccine
  2017-2018 Quadrivalent Inactivated Influenza Vaccine
Period: Overall Study
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Started | 43 | 38
Safety Population | 42 (Added subject randomized to sequential but got simultaneous.) | 38 (Excluded sub. randomized but not vaccinated. Excluded sub. randomized to seq. but got simultaneous.)
Completed | 42 | 38
Not Completed | 1 | 0
Not completed — Randomized but not Vaccinated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Sequential Vaccination Arm: In this study arm, subjects will receive the IIV vaccine during study visit 1. Approximately 21 days later, they will receive the Tdap vaccine during study visit 4.
  Tetanus, Diphtheria, and Pertussis Vaccine
  2016-2017 Quadrivalent Inactivated Influenza Vaccine
  2017-2018 Quadrivalent Inactivated Influenza Vaccine
- Total: Total of all reporting groups
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm | Total
Number analyzed (Participants) | 42 | 38 | 80
Age, Customized [Median (Full Range); unit: Years]
  Maternal Age | 27 [17 to 42] | 25.5 [18 to 39] | 26 [17 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 38 | 80
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 34 | 33 | 67
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 17 | 34
  White | 22 | 17 | 39
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 38 | 80
Recent Tdap Vaccine within 2 years [Count of Participants; unit: Participants] | 5 | 5 | 10
Recent Flu Vaccine within 2 years [Count of Participants; unit: Participants] | 8 | 7 | 15
Gestational Age in Weeks at Visit 1 [Median (Full Range); unit: Weeks] | 29.1 [25.7 to 31.7] | 28 [24.3 to 31.4] | 28.7 [24.3 to 31.7]
Gestational Age in Weeks at Visit 4 [Median (Full Range); unit: Weeks] | 32.6 [29.0 to 36.4] | 31.9 [27.4 to 35.4] | 32.3 [27.4 to 36.4]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Injection-site Reactions Post Tdap and IIV4 Administration
Description: Percentage of injection-site reactions will be compared in simultaneous and sequential groups as determined by self-assessment via memory aid
Time Frame: 8 days post vaccine administration
Population: Safety Population - subjects that were randomized and received the study intervention
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 42 | 38
percentage of participants
  Flu Pain : None: number analyzed (Participants) | 40 | 37
  Flu Pain : None | 47.5 [31.5 to 63.9] | 48.6 [31.9 to 65.6]
  Flu Pain : Mild: number analyzed (Participants) | 40 | 37
  Flu Pain : Mild | 37.5 [22.7 to 54.2] | 45.9 [29.5 to 63.1]
  Flu Pain : Moderate: number analyzed (Participants) | 40 | 37
  Flu Pain : Moderate | 15.0 [5.7 to 29.8] | 5.4 [0.7 to 18.2]
  Flu Pain : Severe: number analyzed (Participants) | 40 | 37
  Flu Pain : Severe | 0 [NA to 8.8] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 9.5] — Cannot estimate lower bound as percentage is 0
  Flu Tenderness : None: number analyzed (Participants) | 40 | 37
  Flu Tenderness : None | 32.5 [18.6 to 49.1] | 54.1 [36.9 to 70.5]
  Flu Tenderness : Mild: number analyzed (Participants) | 40 | 37
  Flu Tenderness : Mild | 55.0 [38.5 to 70.7] | 37.8 [22.5 to 55.2]
  Flu Tenderness : Moderate: number analyzed (Participants) | 40 | 37
  Flu Tenderness : Moderate | 12.5 [4.2 to 26.8] | 8.1 [1.7 to 21.9]
  Flu Tenderness : Severe: number analyzed (Participants) | 40 | 37
  Flu Tenderness : Severe | 0 [NA to 8.8] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 9.5] — Cannot estimate lower bound as percentage is 0
  Tdap Pain : None: number analyzed (Participants) | 40 | 34
  Tdap Pain : None | 55.0 [38.5 to 70.7] | 70.6 [52.5 to 84.9]
  Tdap Pain : Mild: number analyzed (Participants) | 40 | 34
  Tdap Pain : Mild | 30.0 [16.6 to 46.5] | 14.7 [5.0 to 31.1]
  Tdap Pain : Moderate: number analyzed (Participants) | 40 | 34
  Tdap Pain : Moderate | 10.0 [2.8 to 23.7] | 14.7 [5.0 to 31.1]
  Tdap Pain : Severe: number analyzed (Participants) | 40 | 34
  Tdap Pain : Severe | 5.0 [0.6 to 16.9] | 0 [NA to 10.3] — Cannot estimate lower bound as percentage is 0
  Tdap Tenderness : None: number analyzed (Participants) | 40 | 34
  Tdap Tenderness : None | 37.5 [22.7 to 54.2] | 50.0 [32.4 to 67.6]
  Tdap Tenderness : Mild: number analyzed (Participants) | 40 | 34
  Tdap Tenderness : Mild | 37.5 [22.7 to 54.2] | 17.6 [6.8 to 34.5]
  Tdap Tenderness : Moderate: number analyzed (Participants) | 40 | 34
  Tdap Tenderness : Moderate | 22.5 [10.8 to 38.5] | 29.4 [15.1 to 47.5]
  Tdap Tenderness : Severe: number analyzed (Participants) | 40 | 34
  Tdap Tenderness : Severe | 2.5 [0.1 to 13.2] | 2.9 [0.1 to 15.3]
  Flu Redness : None: number analyzed (Participants) | 40 | 37
  Flu Redness : None | 92.5 [79.6 to 98.4] | 83.8 [68.0 to 93.8]
  Flu Redness : Mild: number analyzed (Participants) | 40 | 37
  Flu Redness : Mild | 7.5 [1.6 to 20.4] | 13.5 [4.5 to 28.8]
  Flu Redness : Moderate: number analyzed (Participants) | 40 | 37
  Flu Redness : Moderate | 0 [NA to 8.8] — Cannot estimate lower bound as percentage is 0 | 2.7 [0.7 to 14.2]
  Flu Redness : Severe: number analyzed (Participants) | 40 | 37
  Flu Redness : Severe | 0 [NA to 8.8] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 9.5] — Cannot estimate lower bound as percentage is 0
  Flu Swelling : None: number analyzed (Participants) | 40 | 37
  Flu Swelling : None | 92.5 [79.6 to 98.4] | 89.2 [74.6 to 97.0]
  Flu Swelling : Mild: number analyzed (Participants) | 40 | 37
  Flu Swelling : Mild | 7.5 [1.6 to 20.4] | 8.1 [1.7 to 21.9]
  Flu Swelling : Moderate: number analyzed (Participants) | 40 | 37
  Flu Swelling : Moderate | 0 [NA to 8.8] — Cannot estimate lower bound as percentage is 0 | 2.7 [0.7 to 14.2]
  Flu Swelling : Severe: number analyzed (Participants) | 40 | 37
  Flu Swelling : Severe | 0 [NA to 8.8] — Cannot estimate lower bound as percentage is 0 | 0 [0 to 9.5]
  Tdap Redness : None: number analyzed (Participants) | 40 | 34
  Tdap Redness : None | 85.0 [70.2 to 94.3] | 82.4 [65.5 to 93.2]
  Tdap Redness : Mild: number analyzed (Participants) | 40 | 34
  Tdap Redness : Mild | 15.0 [5.7 to 29.8] | 11.8 [3.3 to 27.5]
  Tdap Redness : Moderate: number analyzed (Participants) | 40 | 34
  Tdap Redness : Moderate | 0 [NA to 8.8] — Cannot estimate lower bound as percentage is 0 | 5.9 [0.7 to 19.7]
  Tdap Redness : Severe: number analyzed (Participants) | 40 | 34
  Tdap Redness : Severe | 0 [NA to 8.8] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 10.3] — Cannot estimate lower bound as percentage is 0
  Tdap Swelling : None: number analyzed (Participants) | 40 | 34
  Tdap Swelling : None | 82.5 [67.2 to 92.7] | 85.3 [68.9 to 95.0]
  Tdap Swelling : Mild: number analyzed (Participants) | 40 | 34
  Tdap Swelling : Mild | 17.5 [7.3 to 32.8] | 11.8 [3.3 to 27.5]
  Tdap Swelling : Moderate: number analyzed (Participants) | 40 | 34
  Tdap Swelling : Moderate | 0 [NA to 8.8] — Cannot estimate lower bound as percentage is 0 | 2.9 [0.1 to 14.2]
  Tdap Swelling : Severe: number analyzed (Participants) | 40 | 34
  Tdap Swelling : Severe | 0 [NA to 8.8] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 10.3] — Cannot estimate lower bound as percentage is 0

2. Primary Outcome: Percentage of Participants With Systemic Reactions Post Tdap and IIV4 Administration - Visit 1
Description: Percentage of systemic reactions will be compared in simultaneous and sequential groups as determined by self-assessment via memory aid
Time Frame: 8 days post vaccine administration
Population: Safety Population - subjects that were randomized and received the study intervention. Participants analyzed include those that provided data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 40 | 37
percentage of participants
  Fever : None | 100.0 [91.2 to 100] | 94.6 [81.8 to 99.3]
  Fever : Mild | 0 [NA to 8.8] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 9.5] — Cannot estimate lower bound as percentage is 0
  Fever : Moderate | 0 [NA to 8.8] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 9.5] — Cannot estimate lower bound as percentage is 0
  Fever : Severe | 0 [NA to 8.8] — Cannot estimate lower bound as percentage is 0 | 5.4 [0.7 to 18.2]
  Abdominal Pain : None | 90.0 [76.3 to 97.2] | 97.3 [85.8 to 99.9]
  Abdominal Pain : Mild | 7.5 [1.6 to 20.4] | 2.7 [0.1 to 14.2]
  Abdominal Pain : Moderate | 2.5 [0.1 to 13.2] | 0 [NA to 9.5] — Cannot estimate lower bound as percentage is 0
  Abdominal Pain : Severe | 0 [NA to 8.8] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 9.5] — Cannot estimate lower bound as percentage is 0
  Body Aches : None | 65.0 [48.3 to 79.4] | 78.4 [61.8 to 90.2]
  Body Aches : Mild | 20.0 [9.1 to 35.6] | 18.9 [8.0 to 35.2]
  Body Aches : Moderate | 15.0 [5.7 to 29.8] | 2.7 [0.1 to 14.2]
  Body Aches : Severe | 0 [NA to 8.8] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 9.5] — Cannot estimate lower bound as percentage is 0
  Body Rash : None | 90.0 [76.3 to 97.2] | 97.3 [85.8 to 99.9]
  Body Rash : Mild | 5.0 [0.6 to 16.9] | 0 [NA to 9.5] — Cannot estimate lower bound as percentage is 0
  Body Rash : Moderate | 2.5 [0.1 to 13.2] | 2.7 [0.1 to 14.2]
  Body Rash : Severe | 2.5 [0.1 to 13.2] | 0 [NA to 9.5] — Cannot estimate lower bound as percentage is 0
  Chills Shivering : None | 90.0 [76.3 to 97.2] | 91.9 [78.1 to 98.3]
  Chills Shivering : Mild | 5.0 [0.6 to 16.9] | 8.1 [1.7 to 21.9]
  Chills Shivering : Moderate | 5.0 [0.6 to 16.9] | 0 [NA to 9.5] — Cannot estimate lower bound as percentage is 0
  Chills Shivering : Severe | 0 [NA to 8.8] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 9.5] — Cannot estimate lower bound as percentage is 0
  Diarrhea : None | 87.5 [73.2 to 95.8] | 89.2 [74.6 to 97.0]
  Diarrhea : Mild | 10.0 [2.8 to 23.7] | 10.8 [3.0 to 25.4]
  Diarrhea : Moderate | 2.5 [0.1 to 13.2] | 0 [NA to 9.5] — Cannot estimate lower bound as percentage is 0
  Diarrhea : Severe | 0 [NA to 8.8] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 9.5] — Cannot estimate lower bound as percentage is 0
  Fatigue : None | 65.0 [48.3 to 79.4] | 78.4 [61.8 to 90.2]
  Fatigue : Mild | 20.0 [9.1 to 35.6] | 16.2 [6.2 to 32.0]
  Fatigue : Moderate | 15.0 [5.7 to 29.8] | 5.4 [0.7 to 18.2]
  Fatigue : Severe | 0 [NA to 8.8] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 9.5] — Cannot estimate lower bound as percentage is 0
  Headache : None | 70.0 [53.5 to 83.4] | 75.7 [58.8 to 88.2]
  Headache : Mild | 15.0 [5.7 to 29.8] | 18.9 [8.0 to 35.2]
  Headache : Moderate | 15.0 [5.7 to 29.8] | 5.4 [0.7 to 18.2]
  Headache : Severe | 0 [NA to 8.8] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 9.5] — Cannot estimate lower bound as percentage is 0
  Joint Pain : None | 82.5 [67.2 to 92.7] | 91.9 [78.1 to 98.3]
  Joint Pain : Mild | 15.0 [5.7 to 29.8] | 2.7 [0.1 to 14.2]
  Joint Pain : Moderate | 2.5 [0.1 to 13.2] | 5.4 [0.7 to 18.2]
  Joint Pain : Severe | 0 [NA to 8.8] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 9.5] — Cannot estimate lower bound as percentage is 0
  Nausea : None | 87.5 [73.2 to 95.8] | 89.2 [74.6 to 97.0]
  Nausea : Mild | 7.5 [1.6 to 20.4] | 10.8 [3.0 to 25.4]
  Nausea : Moderate | 5.0 [0.6 to 16.9] | 0 [NA to 9.5] — Cannot estimate lower bound as percentage is 0
  Nausea : Severe | 0 [NA to 8.8] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 9.5] — Cannot estimate lower bound as percentage is 0
  Vomiting : None | 85.0 [70.2 to 94.3] | 97.3 [85.8 to 99.9]
  Vomiting : Mild | 5.0 [0.6 to 16.9] | 2.7 [0.1 to 14.2]
  Vomiting : Moderate | 10 [2.8 to 23.7] | 0 [NA to 9.5] — Cannot estimate lower bound as percentage is 0
  Vomiting : Severe | 0 [NA to 8.8] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 9.5] — Cannot estimate lower bound as percentage is 0

3. Primary Outcome: Percentage of Participants With Systemic Reactions Post Tdap and IIV4 Administration - Visit 4
Description: as for outcome 2
Time Frame: 8 days post vaccine administration
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 38 | 34
percentage of participants
  Fever : None | 97.4 [86.2 to 99.9] | 100.0 [89.7 to 100.0]
  Fever : Mild | 2.6 [0.1 to 13.8] | 0 [NA to 10.3] — Cannot estimate lower bound as percentage is 0
  Fever : Moderate | 0 [NA to 9.3] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 10.3] — Cannot estimate lower bound as percentage is 0
  Fever : Severe | 0 [NA to 9.3] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 10.3] — Cannot estimate lower bound as percentage is 0
  Abdominal Pain : None | 97.4 [86.2 to 99.9] | 100.0 [89.7 to 100.0]
  Abdominal Pain : Mild | 0 [NA to 9.3] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 10.3] — Cannot estimate lower bound as percentage is 0
  Abdominal Pain : Moderate | 2.6 [0.1 to 13.8] | 0 [NA to 10.3] — Cannot estimate lower bound as percentage is 0
  Abdominal Pain : Severe | 0 [NA to 9.3] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 10.3] — Cannot estimate lower bound as percentage is 0
  Body Aches : None | 92.1 [78.6 to 98.3] | 82.4 [65.5 to 93.2]
  Body Aches : Mild | 0 [NA to 9.3] — Cannot estimate lower bound as percentage is 0 | 11.8 [3.3 to 27.5]
  Body Aches : Moderate | 5.3 [0.6 to 17.7] | 5.9 [0.7 to 19.7]
  Body Aches : Severe | 2.6 [0.1 to 13.8] | 0 [NA to 10.3] — Cannot estimate lower bound as percentage is 0
  Body Rash : None | 100.0 [90.7 to 100.0] | 100.0 [89.7 to 100.0]
  Body Rash : Mild | 0 [NA to 9.3] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 10.3] — Cannot estimate lower bound as percentage is 0
  Body Rash : Moderate | 0 [NA to 9.3] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 10.3] — Cannot estimate lower bound as percentage is 0
  Body Rash : Severe | 0 [NA to 9.3] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 10.3] — Cannot estimate lower bound as percentage is 0
  Chills Shivering : None | 94.7 [82.3 to 99.4] | 97.1 [84.7 to 99.9]
  Chills Shivering : Mild | 5.3 [0.6 to 17.7] | 2.9 [0.1 to 15.3]
  Chills Shivering : Moderate | 0 [NA to 9.3] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 10.3] — Cannot estimate lower bound as percentage is 0
  Chills Shivering : Severe | 0 [NA to 9.3] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 10.3] — Cannot estimate lower bound as percentage is 0
  Diarrhea : None | 97.4 [86.2 to 99.9] | 97.1 [84.7 to 99.9]
  Diarrhea : Mild | 0 [NA to 9.3] — Cannot estimate lower bound as percentage is 0 | 2.9 [0.1 to 15.3]
  Diarrhea : Moderate | 2.6 [0.1 to 13.8] | 0 [NA to 10.3] — Cannot estimate lower bound as percentage is 0
  Diarrhea : Severe | 0 [NA to 9.3] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 10.3] — Cannot estimate lower bound as percentage is 0
  Fatigue : None | 84.2 [68.7 to 94.0] | 85.3 [68.9 to 95.0]
  Fatigue : Mild | 5.3 [0.6 to 17.7] | 11.8 [3.3 to 27.5]
  Fatigue : Moderate | 10.5 [2.9 to 24.8] | 2.9 [0.1 to 15.3]
  Fatigue : Severe | 0 [NA to 9.3] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 10.3] — Cannot estimate lower bound as percentage is 0
  Headache : None | 92.1 [78.6 to 98.3] | 79.4 [62.1 to 91.3]
  Headache : Mild | 2.6 [0.1 to 13.8] | 14.7 [5.0 to 31.1]
  Headache : Moderate | 2.6 [0.1 to 13.8] | 5.9 [0.7 to 19.7]
  Headache : Severe | 2.6 [0.1 to 13.8] | 0 [NA to 10.3] — Cannot estimate lower bound as percentage is 0
  Joint Pain : None | 100.0 [90.7 to 100.0] | 94.1 [80.3 to 99.3]
  Joint Pain : Mild | 0 [NA to 9.3] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 10.3] — Cannot estimate lower bound as percentage is 0
  Joint Pain : Moderate | 0 [NA to 9.3] — Cannot estimate lower bound as percentage is 0 | 5.9 [0.7 to 19.7]
  Joint Pain : Severe | 0 [NA to 9.3] — Cannot estimate lower bound as percentage is 0 | 0 [NA to 10.3] — Cannot estimate lower bound as percentage is 0
  Nausea : None | 94.7 [82.3 to 99.4] | 82.4 [65.5 to 93.2]
  Nausea : Mild | 2.6 [0.1 to 13.8] | 8.8 [1.9 to 23.7]
  Nausea : Moderate | 2.6 [0.1 to 13.8] | 5.9 [0.7 to 19.7]
  Nausea : Severe | 0 [NA to 9.3] — Cannot estimate lower bound as percentage is 0 | 2.9 [0.1 to 15.3]
  Vomiting : None | 94.7 [82.3 to 99.4] | 91.2 [76.3 to 98.1]
  Vomiting : Mild | 5.3 [0.6 to 17.7] | 2.9 [0.1 to 15.3]
  Vomiting : Moderate | 0 [NA to 9.3] — Cannot estimate lower bound as percentage is 0 | 2.9 [0.1 to 15.3]
  Vomiting : Severe | 0 [NA to 9.3] — Cannot estimate lower bound as percentage is 0 | 2.9 [0.1 to 15.3]

4. Primary Outcome: Pertussis Serum Antibody Levels, as Measured by Geometric Mean Titers
Description: Measurement of serum antibody levels to pertussis antigens, in maternal blood pre- and post-vaccination, maternal blood at delivery and infant cord blood obtained at delivery
Time Frame: Pre-vaccination and approximately 21 days post vaccination and at Delivery
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Concentration (IU/mL)
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 42 | 38
Concentration (IU/mL)
  Pre-Vaccination - FHA | 27.5 [18.5 to 41.0] | 37.0 [23.8 to 57.6]
  Pre-Vaccination - FIM | 87.3 [46.9 to 162.4] | 20.8 [10.5 to 41.1]
  Pre-Vaccination - PRN | 44.8 [27.3 to 73.7] | 47.1 [26.4 to 83.9]
  Pre-Vaccination - PT | 7.8 [5.1 to 11.9] | 5.9 [3.5 to 10.1]
  Post-Vaccination - FHA: number analyzed (Participants) | 41 | 38
  Post-Vaccination - FHA | 171.3 [135.0 to 217.7] | 262.1 [201.5 to 341.0]
  Post-Vaccination - FIM: number analyzed (Participants) | 41 | 38
  Post-Vaccination - FIM | 99.9 [55.9 to 178.7] | 19.7 [10.2 to 38.1]
  Post-Vaccination - PRN: number analyzed (Participants) | 41 | 38
  Post-Vaccination - PRN | 242.1 [178.1 to 329.2] | 360.4 [240.8 to 539.4]
  Post-Vaccination - PT: number analyzed (Participants) | 41 | 38
  Post-Vaccination - PT | 37.6 [26.8 to 52.9] | 38.6 [28.4 to 52.3]
  Maternal - FHA: number analyzed (Participants) | 38 | 38
  Maternal - FHA | 118.3 [89.9 to 155.6] | 199.8 [146.7 to 272.1]
  Maternal - FIM: number analyzed (Participants) | 38 | 38
  Maternal - FIM | 81.2 [44.0 to 149.9] | 18.9 [10.3 to 34.9]
  Maternal - PRN: number analyzed (Participants) | 38 | 38
  Maternal - PRN | 174.1 [122 to 248.5] | 297.1 [194.7 to 453.4]
  Maternal - PT: number analyzed (Participants) | 38 | 38
  Maternal - PT | 26.8 [19.3 to 37.4] | 27.9 [19.4 to 40.1]
  Cord Blood - FHA: number analyzed (Participants) | 38 | 35
  Cord Blood - FHA | 182 [137 to 241.8] | 265.6 [195.8 to 360.3]
  Cord Blood - FIM: number analyzed (Participants) | 38 | 35
  Cord Blood - FIM | 122.2 [67.5 to 221.5] | 32.2 [17.5 to 59.4]
  Cord Blood - PRN: number analyzed (Participants) | 38 | 35
  Cord Blood - PRN | 245.4 [171.8 to 350.3] | 352.1 [230.7 to 537.5]
  Cord Blood - PT: number analyzed (Participants) | 38 | 35
  Cord Blood - PT | 46 [32.4 to 65.2] | 43.4 [29.8 to 62.3]

5. Primary Outcome: Percentage of Subjects With Seroprotection as Determined by Diphtheria Serum Antibody Levels (Defined as ≥ 0.1 IU/mL)
Description: Measurement of serum antibody levels to diphtheria toxoids, in maternal blood pre- and post-vaccination, maternal blood at delivery and infant cord blood obtained at delivery
Time Frame: Pre vaccination and approximately 21 days post vaccination and at Delivery
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 41 | 37
percentage of participants
  Pre-Vaccination: number analyzed (Participants) | 40 | 37
  Pre-Vaccination | 62.5 [45.8 to 77.3] | 76.3 [59.8 to 88.6]
  Post-Vaccination | 92.7 [80.1 to 98.5] | 100 [90.5 to NA] — Cannot be estimated - value is already 100%
  Maternal Blood: number analyzed (Participants) | 38 | 37
  Maternal Blood | 92.1 [78.6 to 98.3] | 100.0 [90.5 to NA] — Cannot be estimated - value is already 100%
  Cord Blood: number analyzed (Participants) | 38 | 32
  Cord Blood | 94.7 [82.3 to 99.4] | 100.0 [89.1 to NA] — Cannot be estimated - value is already 100%

6. Primary Outcome: Percentage of Subjects With Seroprotection as Determined by Tetanus Serum Antibody Levels (Defined as ≥ 0.1 IU/mL)
Description: Measurement of serum antibody levels to tetanus toxoids, in maternal blood pre- and post-vaccination, maternal blood at delivery and infant cord blood obtained at delivery
Time Frame: 21 days post vaccination
Population: Safety Population - all subjects receiving the study intervention. Participants analyzed include those that provided data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 41 | 38
percentage of participants
  Pre-Vaccination: number analyzed (Participants) | 40 | 38
  Pre-Vaccination | 82.5 [67.2 to 92.7] | 84.2 [68.7 to 94.0]
  Post-Vaccination: number analyzed (Participants) | 41 | 37
  Post-Vaccination | 97.6 [87.1 to 99.9] | 100 [90.5 to NA] — Cannot be estimated - value is already 100%
  Maternal Blood: number analyzed (Participants) | 38 | 37
  Maternal Blood | 100.0 [90.7 to NA] — Cannot be estimated - value is already 100% | 97.3 [85.8 to 99.9]
  Cord Blood: number analyzed (Participants) | 38 | 32
  Cord Blood | 100.0 [90.7 to NA] — Cannot be estimated - value is already 100% | 100.0 [89.1 to NA] — Cannot be estimated - value is already 100%

7. Primary Outcome: Percentage of Subjects With Seroprotection as Determined by Influenza Serum Antibody Levels (≥1:40) (Pre- and Post-immunization) and Seroconversion (4-fold Rise From Baseline or a Change From <1:10 to ≥1:40) )
Description: Measurement of serum antibody levels to influenza antigens in maternal blood and infant cord blood obtained at delivery
Time Frame: Pre and 21 days post vaccination and at Delivery
Population: Safety Population - subjects receiving the study intervention. Participants analyzed include those that provided data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 41 | 38
percentage of participants
  A/H1N1: Pre-Vaccination Seroprotection | 58.5 [42.1 to 73.7] | 71.1 [54.1 to 84.6]
  A/H1N1: Post-Vaccination Seroprotection | 90.2 [76.9 to 97.3] | 94.7 [82.3 to 99.4]
  A/H1N1: Seroconversion | 39.0 [24.2 to 55.5] | 50.0 [33.4 to 66.6]
  A/H3N2: Pre-Vaccination Seroprotection | 53.7 [37.4 to 69.3] | 60.5 [43.4 to 76.0]
  A/H3N2: Post-Vaccination Seroprotection | 95.1 [83.5 to 99.4] | 92.1 [78.6 to 98.3]
  A/H3N2: Seroconversion | 63.4 [46.9 to 77.9] | 65.8 [48.6 to 80.4]
  B/Brisbane: Pre-Vaccination Seroprotection | 14.6 [5.6 to 29.2] | 13.2 [4.4 to 28.1]
  B/Brisbane: Post-Vaccination Seroprotection | 63.4 [46.9 to 77.9] | 63.2 [46.0 to 78.2]
  B/Brisbane: Seroconversion | 53.7 [37.4 to 69.3] | 50.0 [33.4 to 66.6]
  B/Phuket: Pre-Vaccination Seroprotection | 29.3 [16.1 to 45.5] | 47.4 [31.0 to 64.2]
  B/Phuket: Post-Vaccination Seroprotection | 78.0 [62.4 to 89.4] | 81.6 [65.7 to 92.3]
  B/Phuket: Seroconversion | 58.5 [42.1 to 73.7] | 42.1 [26.3 to 59.2]
  A/H1N1: Maternal Seroprotection: number analyzed (Participants) | 38 | 37
  A/H1N1: Maternal Seroprotection | 89.5 [75.2 to 97.1] | 94.6 [81.8 to 99.3]
  A/H1N1: Cord Blood Seroprotection: number analyzed (Participants) | 38 | 32
  A/H1N1: Cord Blood Seroprotection | 97.4 [86.2 to 99.9] | 93.8 [79.2 to 99.2]
  A/H3N2: Maternal Seroprotection: number analyzed (Participants) | 38 | 37
  A/H3N2: Maternal Seroprotection | 92.1 [78.6 to 98.3] | 94.6 [81.8 to 99.3]
  A/H3N2: Cord Blood Seroprotection: number analyzed (Participants) | 38 | 32
  A/H3N2: Cord Blood Seroprotection | 100.0 [90.7 to NA] — Cannot be estimated - value is already 100% | 100.0 [89.1 to NA] — Cannot be estimated - value is already 100%
  B/Brisbane: Maternal Seroprotection: number analyzed (Participants) | 38 | 37
  B/Brisbane: Maternal Seroprotection | 42.1 [26.3 to 59.2] | 51.4 [34.4 to 68.1]
  B/Brisbane: Cord Blood Seroprotection: number analyzed (Participants) | 38 | 32
  B/Brisbane: Cord Blood Seroprotection | 76.3 [59.8 to 88.6] | 78.1 [60.0 to 90.7]
  B/Phuket: Maternal Seroprotection: number analyzed (Participants) | 38 | 37
  B/Phuket: Maternal Seroprotection | 73.7 [56.9 to 86.6] | 67.6 [50.2 to 82.0]
  B/Phuket: Cord Blood Seroprotection: number analyzed (Participants) | 38 | 32
  B/Phuket: Cord Blood Seroprotection | 81.6 [65.7 to 92.3] | 87.5 [71.0 to 96.5]

8. Primary Outcome: Percentage of Subjects Recruited Enrollment Period
Description: Percentage of subjects recruited during 4 month enrollment period
Time Frame: Approximately 1 year
Population: All subjects recruited and enrolled in the study
Measure: Number; unit: percentage of participants
Groups:
- Recruited Subjects: In the study arm, this includes all subjects that were recruited and enrolled into the study.
Arm/Group | Recruited Subjects
Number analyzed (Participants) | 81
percentage of participants | 100.0

9. Primary Outcome: Feasibility as Measured by Participant Retention (Percentage of Participants Who Complete All Visits)
Description: Percentage of participants that completed all in-person and delivery visits
Time Frame: Approximately 1 year
Population: Safety Population - subjects randomized and received study intervention
Measure: Number; unit: percentage of participants
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 42 | 38
percentage of participants | 98.6 | 97.7

10. Primary Outcome: Feasibility Reported as Percentage of Reactogenicity Data Collected
Description: Percentage of reactogenicity data days reported (days reported / total possible days)
Time Frame: Approximately 1 year
Population: Safety Population - subjects randomized and received study intervention
Measure: Number; unit: percentage of days
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 42 | 38
percentage of days | 92.6 | 93.1

11. Primary Outcome: Feasibility Reported as Percentage of Adequate Biospecimens Collected
Description: Percentage of samples collected (sample timepoints collected / total possible sample timepoints)
Time Frame: Approximately 1 year
Population: Safety Population - subjects randomized and received study intervention
Measure: Number; unit: percentage of samples
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 42 | 38
percentage of samples | 94.0 | 95.4

12. Primary Outcome: Feasibility Reported as Percentage of Timely Collected Biospecimens
Description: Timeliness is defined as collected within the visit window
Time Frame: Approximately 1 year
Population: Safety Population - subjects randomized and received study intervention
Measure: Number; unit: percentage of samples
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 42 | 38
percentage of samples | 94.0 | 95.4

13. Secondary Outcome: Number of Participants With Adverse Maternal Outcomes
Description: The number of participants with adverse maternal outcomes at delivery. Missing data is data not collected or unavailable.
Time Frame: Up to the 6-week postpartum visit
Population: Safety Population - subjects randomized and received study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 42 | 38
Participants
  Pre-term Birth (<37 weeks): Yes | 3 | 0
  Pre-term Birth (<37 weeks): No | 38 | 37
  Pre-term Birth (<37 weeks): Missing | 1 | 1
  Gestational Diabetes: Yes | 6 | 3
  Gestational Diabetes: No | 35 | 35
  Gestational Diabetes: Missing | 1 | 0
  Gestational Hypertension: Yes | 5 | 7
  Gestational Hypertension: No | 36 | 31
  Gestational Hypertension: Missing | 1 | 0
  Preeclampsia: Yes | 3 | 1
  Preeclampsia: No | 38 | 37
  Preeclampsia: Missing | 1 | 0
  Severe Preeclampsia/HELLP: Yes | 1 | 0
  Severe Preeclampsia/HELLP: No | 40 | 38
  Severe Preeclampsia/HELLP: Missing | 1 | 0

14. Secondary Outcome: Number of Participants With Adverse Infant Outcomes Based on Medical Record Review
Description: Number of participants with adverse infant outcomes. Missing data is data not collected or unavailable.
Time Frame: approximately 2 months
Population: Safety Population - subjects randomized and received study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 42 | 38
Participants
  Small Gestational Age (SGA): Olsen et al.: Yes | 2 | 4
  Small Gestational Age (SGA): Olsen et al.: No | 40 | 34
  Small Gestational Age (SGA): Olsen et al.: Missing | 0 | 0
  Neonatal Death: Yes | 0 | 0
  Neonatal Death: No | 41 | 38
  Neonatal Death: Missing | 1 | 0
  Hypoglycemia: Yes | 0 | 1
  Hypoglycemia: No | 41 | 37
  Hypoglycemia: Missing | 1 | 0
  Respiratory: Yes | 0 | 1
  Respiratory: No | 41 | 37
  Respiratory: Missing | 1 | 0
  Jaundice Requiring Phototherapy: Yes | 1 | 1
  Jaundice Requiring Phototherapy: No | 40 | 37
  Jaundice Requiring Phototherapy: Missing | 1 | 0
  Transient Tachypnea: Yes | 1 | 0
  Transient Tachypnea: No | 40 | 38
  Transient Tachypnea: Missing | 1 | 0
  Hematological: Yes | 0 | 2
  Hematological: No | 41 | 36
  Hematological: Missing | 1 | 0
  Sepsis/Rule out Infection: Yes | 1 | 1
  Sepsis/Rule out Infection: No | 40 | 37
  Sepsis/Rule out Infection: Missing | 1 | 0
  Low Birth Weight (< 2500 g): Yes | 3 | 2
  Low Birth Weight (< 2500 g): No | 38 | 35
  Low Birth Weight (< 2500 g): Missing | 1 | 1

15. Secondary Outcome: Percentage of Participants With Clinical Chorioamnionitis
Description: Percentage of participants with clinical chorioamnionitis
Time Frame: at the time of delivery
Population: Safety Population - subjects randomized and receiving study intervention
Measure: Number; unit: percentage of participants
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 42 | 38
percentage of participants | 0.0 | 0.0

16. Secondary Outcome: Percentage of Participants With Histologic Chorioamnionitis on Surgical Pathology Examination of Placental Tissue
Description: Percentage of participants with histologic chorioamnionitis on surgical pathology examination of placental tissue
Time Frame: after delivery, approximately up to 2 weeks
Population: Safety Population - subjects randomized and received study intervention
Measure: Number; unit: percentage of participants
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 42 | 38
percentage of participants | 19.0 | 15.8

17. Secondary Outcome: Feasibility as Measured by Percentage of Blood Samples in Testable Condition
Description: Percentage of blood samples received in testable condition (sufficient volume and quality)
Time Frame: Approximately 1 year
Population: Safety Population - subjects randomized and received study intervention
Measure: Number; unit: percentage of samples
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 42 | 38
percentage of samples | 100.0 | 100.0

18. Secondary Outcome: Feasibility as Measured by Percentage of Blood Samples in With Sufficient Volume for Testing
Description: Percentage of blood samples received with sufficient volume for testing
Time Frame: Approximately 1 year
Population: Safety Population - subjects randomized and received study intervention
Measure: Number; unit: percentage of samples
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 42 | 38
percentage of samples | 100.0 | 100.0

19. Secondary Outcome: Feasibility as Measured by Percentage of Testable Blood Samples Completed
Description: Percentage of testable (sufficient volume and quality) blood samples completed
Time Frame: Approximately 1 year
Population: Safety Population - subjects randomized and received study intervention
Measure: Number; unit: percentage of samples
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
Number analyzed (Participants) | 42 | 38
percentage of samples | 100.0 | 100.0

ADVERSE EVENTS:
Time Frame: Adverse events and SAEs are captured up to 8 days post vaccination. Subjects are followed for SAEs up to the 6-week postpartum visit. Significant infant complications or SAEs identified during the delivery visit will be followed up to the 2-month well child visit.
Description: All-cause mortality, serious adverse events, and other AEs exceeding a frequency threshold of 5% were collected and reported.
Arm/Group | Simultaneous Vaccination Arm | Sequential Vaccination Arm
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/38
Serious Adverse Events (participants affected / at risk) | 1/42 | 0/38
Other Adverse Events (participants affected / at risk) | 2/42 | 2/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simultaneous Vaccination Arm (N=42) | Sequential Vaccination Arm (N=38)
Uterine Rupture (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Uterine rupture with cesarean delivery and hysterectomy. Assessed as unrelated to vaccine.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simultaneous Vaccination Arm (N=42) | Sequential Vaccination Arm (N=38)
Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Headaches (General disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT02783170/Prot_SAP_000.pdf
  • Informed Consent Form (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT02783170/ICF_001.pdf